CLINICAL TRIAL: NCT01459926
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Assess the Safety and Efficacy of TD-1211 in Subjects With Opioid-Induced Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0084
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Opioid Induced Constipation
Keywords: Opioid induced constipation; OIC; Constipation; Opioid side effects; Morphine induced constipation; Opioid therapy
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation | interventions — 3-(8-(2-(cyclohexylmethyl(2,3-dihydroxypropionyl)amino)ethyl)-8-azabicyclo(3.2.1)oct-3-yl)benzamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose 1 (Experimental)
  Interventions: Drug: TD-1211
- Dose 2 (Experimental)
  Interventions: Drug: TD-1211
- Dose 3 (Experimental)
  Interventions: Drug: TD-1211
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-1211 — once daily
  Arms: Dose 1
Drug: TD-1211 — Once daily
  Arms: Dose 2
Drug: TD-1211 — Once daily
  Arms: Dose 3
Drug: Placebo — Once daily
  Arms: Placebo

SUMMARY:
A Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Assess the Safety and Efficacy of TD-1211 in Subjects with Opioid-Induced Constipation

ELIGIBILITY:
Inclusion Criteria:

* History of constipation with onset after initiation of opioid therapy
* Self-reported OIC of approximately 3 spontaneous bowel movements (SBMs) per week or less for each week over at least the previous two week period
* Have used chronic opioids with a total daily dose ≥30 mg of morphine equivalent units (MEU, Appendix 7) for the 12 weeks preceding the Screening Visit. Subjects should have used a stable daily regimen of opioids for at least the 2 weeks preceding the Screening Visit
* Willing to stop all laxatives and other bowel regimens with the exception of bisacodyl/enema treatment allowed per protocol throughout the OIC confirmation, treatment, and follow-up periods

Exclusion Criteria:

* Have participated in a clinical trial of an investigational drug or medical device within 30 days prior to Screening
* Have any condition that may affect drug absorption, (e.g., previous GI surgery)
* Any other condition which, in the opinion of the investigator, could confound or interfere with evaluation of safety or tolerability of the investigational drug, or prevent compliance with the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the weekly average CSBMs over Weeks 2 to 5 of treatment | Between weeks 2 and 5

SECONDARY OUTCOMES:
Change from baseline in the weekly SBM frequency in the last week of treatment | baseline and 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- G and L Research, LLC, Foley, Alabama, United States